CLINICAL TRIAL: NCT02752737
Title: Cryo Global Registry, a Part of the Medtronic Cardiac Ablation Post-Market Study Platform
Brief Title: Cryo Global Registry
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: Cryo Global Registry
Record Dates: First submitted 2016-04-25; First posted 2016-04-27 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Cryo Global Registry a prospective, global, multi-center, observational Post-Market Registry

DETAILED DESCRIPTION:
The Cryo Global Registry is a prospective, global, multi-center, observational post-market registry (PMR). The purpose of this study is to evaluate and describe clinical performance and safety data in a broad patient population treated with a commercially available Arctic Front™ Family of Cardiac Cryoablation Catheters (hereafter referred to as "Arctic Front™ Cardiac Cryoablation Catheter System"). The cryoballoon ablation(CBA) procedure will be performed according to routine hospital practice. The study is expected to have a 24 month enrollment period. The follow up period is intended to align with standard practice and subjects will be followed for a minimum of 12 months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age or minimum age as required by local regulations
* Planned procedure using commercially available Arctic Front™ Cardiac Cryoablation Catheter
* Willing to comply with study requirements and give informed consent (defined as legally effective, documented confirmation of a subject's voluntary agreement to participate in this clinical study) or authorization per institution and geographical requirements

Exclusion Criteria:

* Subject is enrolled in a concurrent study that has not been approved for concurrent enrollment by the global study manager
* Subject with exclusion criteria required by local law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years or older with a planned procedure using commercially available Arctic Front™ Cardiac Cryoablation Catheter.
Sampling Method: Non-Probability Sample
Enrollment: 5385 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
Freedom from Atrial Fibrillation (AF) Recurrence at 12 Months | 12 Months
  Estimate the 12 month freedom from AF recurrence using the Arctic Front™ Cardiac Cryoablation Catheter System
Freedom from Atrial Arrhythmia at 12 Months | 12 Months
  Estimate the 12 month freedom from AF / Atrial Flutter (AFL)/ Atrial Tachycardia (AT) using the Arctic Front™ Cardiac Cryoablation Catheter System.
Freedom from Arrythmias at 12 months | 12 Months
  Estimate the 12-month freedom from arrythmias treated using the Freezor™ Family of Cardiac Cryoablation Catheters.
Freedom from Device / Procedure Related Adverse Events | 12 Months
  Estimate device and procedure-related adverse events for cryoablation using the Arctic Front™ Cardiac Cryoablation Catheter System through 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Khaldoun Tarakji, MD, Study Director — Medtronic CAS Chief Medical Officer
Locations (161):
- United States (6):
  - Carle Foundation Hospital, Urbana, Illinois
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - The Lindner Research Center, Cincinnati, Ohio
  - Doylestown Health Cardiology, Doylestown, Pennsylvania
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Texas Health Research & Education Institute, Dallas, Texas
- Argentina (3):
  - Instituto Cardiovascular de Buenos Aires (ICBA), Buenos Aires
  - Institituo Cardiovascular Buenos Aires (ICBA), Buenos Aires
  - Hospital Universitario Fundación Favaloro, Buenos Aires
- Kepler Universitätsklinikum Med Campus III., Linz, Austria
- Belgium (2):
  - Centre Hospitalier Régional de la Citadelle, Liège, Liege
  - Onze-Lieve-Vrouwziekenhuis-Campus Aalst, Aalst
- Gleneagles Jerudong Park Medical Centre, Bandar Seri Begawan, Brunei, Brunei
- Clínica Dávila, Santiago, Chile
- China (6):
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Fuwai Hospital Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing
  - West China Hospital of Sichuan University, Chengdu
  - Shanghai Tenth People's Hospital, Shanghai
  - Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai
  - Tianjin Chest Hospital, Tianjin
- Colombia (2):
  - Fundacion Clinica Shaio, Bogotá
  - Clinica Ces, Medellín
- Nemocnice Na Homolce, Prague, Czechia
- Germany (13):
  - Märkische Gesundheitsholding GmbH & Co. KG - Klinikum Lüdenscheid, Lüdenscheid, North Rhine-Westphalia
  - Herz- und Gefässzentrum Bad Bevensen, Bad Bevensen
  - Segeberger Kliniken GmbH - Herzzentrum, Bad Segeberg
  - Sana Klinikum Lichtenberg, Berlin
  - Städtische Kliniken Bielefeld, Bielefeld
  - Klinikum Coburg GmbH, Coburg
  - St. Vinzenz-Hospital Köln, Cologne
  - Cardioangiologisches Centrum Bethanien, Frankfurt
  - Klinikum Lüdenscheid, Lüdenscheid
  - Kliniken Maria Hilf GmbH Mönchengladbach - Krankenhaus St. Franziskus, Mönchengladbach
  - Städtische Kliniken München GmbH - Klinikum Bogenhausen, München
  - Oberschwaben-Klinik GmbH - Krankenhaus St. Elisabeth, Ravensburg
  - St. Josephs Hospital Wiesbaden, Wiesbaden
- Hellenic Airforce 251 General Hospital, Athens, Greece
- Hungary (2):
  - Gottsegen György Országos Kardiológiai Intézet, Budapest
  - Debreceni Egyetem, Debrecen
- Landspitali - National Hospital of Iceland, Reykjavik, Iceland, Iceland
- India (6):
  - Aster Medcity, Kochi, Kerala
  - Sree Chitra Tirunal Institute for Medical Sciences & Technology, Thiruvananthapuram, Kerala
  - Eternal Hospital, Jaipur, Rajasthan
  - Apollo Hospital (Chennai), Chennai, Tamil Nadu
  - Aig Hospital, Hyderabad
  - Max Super Speciality Hospital, New Delhi
- National Cardiovascular Center Harapan Kita, Jakarta, Indonesia
- Italy (4):
  - Humanitas Mater Domini, Castellanza
  - Fondazione IRCCS Policlinico San, Pavia
  - Ospedale S. Maria della Misericordia, Perugia
  - Azienda Ospedaliero-Universitaria Pisana - Stabilimento di Cisanello, Pisa
- Japan (61):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Japanese Red Cross Nagoya Daini Hospital, Nagoya, Aichi-ken
  - Fukuoka Sanno Hospital, Fukuoka, Fukuoka
  - Ogaki Municipal Hospital, Ōgaki, Gifu
  - Hiroshima City Hospital, Hiroshima, Hiroshima
  - Hiroshima Prefectural Hospital, Hiroshima, Hiroshima
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Hokkaido Ohno Memorial Hospital, Sapporo, Hokkaido
  - Caress Sapporo Hokko Memorial Hospital, Sapporo, Hokkaido
  - Tsuchiura Kyodo General Hospital, Tsuchiura, Ibaraki
  - Tokai University Hospital, Isehara, Kanagawa
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - Japanese Red Cross Wakayama Medical Center, Wakayama, Kansai
  - Miyazaki Medical Association Hospital, Miyazaki, Miyazaki
  - Sakurabashi Watanabe Hospital, Osaka, Osaka
  - Osaka Rosai Hospital, Sakai, Osaka
  - Osaka General Medical Center, Sumiyoshi-ku, Osaka
  - Tokyo University Hospital, Bunkyo-Ku, Tokyo
  - Sakakibara Heart Institute, Fuchū, Tokyo
  - Hyogo Prefectural Amagasaki General Medical Center, Amagasaki
  - Kansai Rosai Hospital, Amagasaki
  - Anjo Kosei Hospital, Anjo
  - Tokyo Medical and Dental University, Medical Hospital, Bunkyō City
  - Nippon Medical School Hospital, Bunkyō City
  - Chiba University Hospital, Chiba
  - Tokai University Hachioji Hospital, Hachiōji
  - Saitama Medical University International Medical Center, Hidaka
  - Hirosaki University Hospital, Hirosaki
  - Hiroshima City Hospital, Hiroshima
  - Kanazawa University Hospital, Ishikawa
  - Nihon University Itabashi Hospital, Itabashi-ku
  - National Hospital Organization Kagoshima MC, Kagoshima
  - Kokura Kinen Hospital, Kitakyushu
  - Kobe City Medical Center General Hospital, Kobe
  - Dokkyo Medical University Saitama Medical Center, Koshigaya
  - Saiseikai Kumamoto Hospital, Kumamoto
  - Kyoto University Hospital, Kyoto
  - The Jikei University School of Medicine Hospital, Minatoku
  - Kyorin University Hospital, Mitaka
  - Mie Heart Center, Miwa
  - Nagoya City University East Medical Center, Nagoya
  - Kochi Medical School Hospital, Nankoku
  - Kurashiki Central Hospital, Okayama
  - Kindai University Hospital, Ōsaka-sayama
  - Toho University Omori Medical Center, Ōta-ku
  - Kitasato University Hospital, Sagamihara
  - Japanese Red Cross Saitama Hospital, Saitama
  - Sendai City Hospital, Sendai
  - Jichi Medical University Hospital, Shimotsuke-shi
  - National Cerebral and Cardiovascular Center, Suita
  - Tenri Hospital, Tenri
  - Showa University Toyosu Hospital, Tokyo
  - Tokyo Medical Center, Tokyo
  - Tokyo Metropolitan Hiroo Hospital, Tokyo
  - Toyama Prefectural Central Hospital, Toyama
  - Fujita Health University Hospital, Toyoake
  - University of Tsukuba Hospital, Tsukuba
  - Yamagata University Hospital, Yamagata
  - Yokkaichi Municipal Hospital, Yokkaichi
  - Yokohama City Minato Red Cross Hospital, Yokohama
  - University of Fukui Hospital, Yoshida
- National Research Cardiac Surgery Center, Astana, Kazakhstan
- Kuwait (2):
  - Salman Al Abdallah Al Dabbous Cardiac Center (DCC) - Al Adan Hospital, Al Ahmadi
  - Chest Diseases Hospital, Kuwait City
- Malaysia (4):
  - Cardiac Vascular Sentral Kuala Lumpur (CVSKL), Kuala Lumpur, Malaysia
  - Sarawak Heart Centre, Kuching, Sarawak
  - Hospital Serdang, Sepang, Selangor
  - Institut Jantung Negara, Kuala Lumpur
- Mexico (3):
  - Hospital Angeles Lomas, Huixquilucan, State of Mexico
  - Centro Médico Nacional Siglo XXI, Mexico City
  - Hospital San Angel Inn Universidad, México
- The Royal Hospital, Muscat, Oman
- Philippines (2):
  - Saint Lukes Medical Center (SLMC), City of Taguig, National Capital Region
  - The Medical City, Pasig, National Capital Region
- Poland (4):
  - Spital Wojewodzki nr 2, Rzeszów, Poland
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II, Krakow
  - Centralny Szpital Kliniczny Uniwersytetu Medycznego w Łodzi, Lodz
  - Kliniczny Szpital Wojewódzki Nr 2 im. Św. Jadwigi Królowej w Rzeszowie, Rzeszów
- Centro hospitalar Vila Nova de Gaia/Espinho-Unidade I, Vila Nova de Gaia, Portugal
- Russia (3):
  - Russian Scientific Center of Surgery by B.V. Petrovskiy, RAMN, Moscow
  - Tomsk National Research Medical Center of the Russian Academy of Sciences, Tomsk
  - State Budgetary Healthcare Institution of Sverdlovsk region for "Sverdlovsk Regional Clinical Hospital #1", Yekaterinburg
- King Fahad Medical City (KFMC), Riyadh, Saudi Arabia
- Institute for Cardiovascular Disease (ICVD) Dedinje, Belgrade, Serbia, Serbia
- Singapore (2):
  - National University Hospital, Singapore
  - National Heart Centre Singapore, Singapore
- Slovakia (3):
  - Stredoslovensky Ustav Srdcovych a Cievnych Chorob a.s, Banská Bystrica
  - Narodny ustav srdcovych a cievnych chorob, a.s. (NUSCH), Bratislava
  - Vychodoslovensky ustav srdcovych a cievnych chorob, a.s., Košice
- South Africa (2):
  - Netcare Sunninghill Hospital, Johannesburg
  - Busamed Gateway Hospital, Umhlanga
- South Korea (3):
  - Seoul National University Bundang Hospital, Seoul, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Seoul
  - Samsung Medical Center, Seoul
- Hospital Universitario Moncloa, Madrid, Spain
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- Taiwan (4):
  - Taichung Veterans General Hospital, Taichung, Taiwan
  - Mackay Memorial Hospital, Taipei, Taiwan
  - Cheng-Hsin General Hospital, Taipei, Taiwan
  - Taipei Veterans General Hospital, Taipei
- Thailand (3):
  - Siriraj Hospital, Bangkok, Thailand
  - Phramongkutklao Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
- United Arab Emirates (2):
  - Cleveland Clinic Abu Dhabi, Abu Dhabi
  - Sheikh Khalifa Medical City, Abu Dhabi
- United Kingdom (5):
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust - Freeman Hospital, Newcastle upon Tyne, United Kingdom
  - Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool
  - St George's University Hospitals - NHS Trust, London
  - St. George's Hospital-NHS Trust, London
  - St. Bartholomew's Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdrakhmanov A, Nuralinov O, Rashbayeva G, Tursunbekov A, Bagibayev S, Bakytzhanuly A, Yessilbayev Z, Chinybayeva A, Abdrakhmanova Z, Salustri A, Suleymen Z, Kirkimbayeva R. Cryoballoon ablation for the treatment of atrial fibrillation in Kazakhstan: One year outcome from the Cryo Global Registry. Indian Pacing Electrophysiol J. 2025 Sep-Oct;25(5):294-301. doi: 10.1016/j.ipej.2025.06.008. Epub 2025 Jun 20. PMID 40545038
- [Derived] Khelae SK, Chun KRJ, Drephal C, Scazzuso F, Kueffer FJ, van Bragt KA, Lawrenz T, Todd D, Ptaszynski P, Foldesi C. Real-world sex differences in healthcare utilization after cryoballoon ablation: 2-year outcomes from the Cryo Global Registry. Front Cardiovasc Med. 2025 Jun 3;12:1549002. doi: 10.3389/fcvm.2025.1549002. eCollection 2025. PMID 40529551
- [Derived] Lawin D, Stellbrink C, Chun KJ, Li CH, van Bragt KA, Kueffer F, Selma JM, Oh IY, Herzet JM, Nitta J, Chang TY, Lawrenz T. Impact of atrial fibrillation diagnosis-to-ablation time on 24-month efficacy and safety outcomes in the Cryo Global Registry. Europace. 2025 Feb 5;27(2):euaf008. doi: 10.1093/europace/euaf008. PMID 39836630
- [Derived] Ahn H, Lim HE, On YK, Selma JM, Kueffer FJ, van Bragt KA, Obidigbo V, Oh IY. Long-term Outcome of Cryoballoon Ablation in Korean Patients With Atrial Fibrillation: Real-World Experience From the Cryo Global Registry. Korean Circ J. 2024 Oct;54(10):619-633. doi: 10.4070/kcj.2024.0044. Epub 2024 Jun 10. PMID 38956935
- [Derived] Lawin D, Lawrenz T, Chun KRJ, Lim HE, Obidigbo V, Selma JM, Peytchev P, Nguyen DQ, Foldesi C, Stellbrink C; the Cryo AF Global Registry Investigators. Cryoballoon ablation of atrial fibrillation in octogenarians: one year outcomes from the cryo global registry. J Interv Card Electrophysiol. 2024 Sep;67(6):1341-1351. doi: 10.1007/s10840-023-01680-z. Epub 2023 Dec 12. PMID 38082096
- [Derived] Scazzuso F, Ptaszynski P, Kaczmarek K, Chun KRJ, Khelae SK, Foldesi C, Obidigbo V, van Bragt KA, On YK, Al-Kandari F, Okumura K; Cryo Global Registry Investigators. Regional variations in patient selection and procedural characteristics for cryoballoon ablation of atrial fibrillation in the cryo global registry. J Interv Card Electrophysiol. 2024 Apr;67(3):493-501. doi: 10.1007/s10840-023-01582-0. Epub 2023 Jul 28. PMID 37505337
- [Derived] Zucchelli G, Chun KRJ, Khelae SK, Foldesi C, Kueffer FJ, van Bragt KA, Scazzuso F, On YK, Al-Kandari F, Okumura K; Cryo Global Registry Investigators. Impact of first-line cryoablation for atrial fibrillation on healthcare utilization, arrhythmia disease burden and efficacy outcomes: real-world evidence from the Cryo Global Registry. J Interv Card Electrophysiol. 2023 Apr;66(3):711-722. doi: 10.1007/s10840-022-01388-6. Epub 2022 Nov 4. PMID 36331681
- [Derived] Lim HE, Oh IY, Kueffer FJ, van Bragt KA, On YK. Cryoballoon Catheter Ablation in Korean Patients With Paroxysmal and Persistent Atrial Fibrillation: One Year Outcome From the Cryo Global Registry. Korean Circ J. 2022 Oct;52(10):755-767. doi: 10.4070/kcj.2022.0127. Epub 2022 Aug 12. PMID 36097833
- [Derived] Rordorf R, Scazzuso F, Chun KRJ, Khelae SK, Kueffer FJ, Braegelmann KM, Okumura K, Al-Kandari F, On YK, Foldesi C; Cryo AF Global Registry Investigators. Cryoballoon Ablation for the Treatment of Atrial Fibrillation in Patients With Concomitant Heart Failure and Either Reduced or Preserved Left Ventricular Ejection Fraction: Results From the Cryo AF Global Registry. J Am Heart Assoc. 2021 Dec 21;10(24):e021323. doi: 10.1161/JAHA.121.021323. Epub 2021 Dec 10. PMID 34889108